CLINICAL TRIAL: NCT01492426
Title: A Phase 3 Evaluation of BMS-790052 (Daclatasvir) Compared With Telaprevir in Combination With Peginterferon Alfa-2a and Ribavirin in Treatment-Naive Patients With Chronic Hepatitis C
Brief Title: Study Comparing Daclatasvir (BMS-790052) With Telaprevir Combined With Peginterferon Alfa-2a and Ribavirin in Patients With Chronic Hepatitis C Virus Infection
Acronym: COMMAND-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI444-052; 2011-004237-14 (EudraCT Number)
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Results first posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-04

CONDITIONS: Hepatitis C
Keywords: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; telaprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daclatasvir + Peginterferon alfa-2a + Ribavirin (Experimental)
  Interventions: Drug: Daclatasvir; Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Telaprevir + Peginterferon alfa-2a + Ribavirin (Experimental)
  Interventions: Drug: Telaprevir; Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Daclatasvir — Film-coated tablet, oral, 60 mg, once daily, 24 weeks
  Other Names: BMS-790052
  Arms: Daclatasvir + Peginterferon alfa-2a + Ribavirin
Drug: Telaprevir — Film-coated tablet, oral, 750 mg, 3 times daily
  Other Names: Incivek®
  Arms: Telaprevir + Peginterferon alfa-2a + Ribavirin
Drug: Peginterferon alfa-2a — Solution for injection, subcutaneous injection, 180 μg, weekly
  Other Names: Pegasys®
Drug: Ribavirin — Film-coated tablet, oral, in a body weight stratified dose range of 1000-1200 mg per day
  Other Names: Copegus®

SUMMARY:
The purpose of this study is to compare the effectiveness of BMS-790052 (Daclatasvir) and Telaprevir when given in combination with Peginterferon alfa-2a and Ribavirin in genotype 1b patients

DETAILED DESCRIPTION:
Allocation: Randomized Stratified

ELIGIBILITY:
Key Inclusion Criteria:

* Participants chronically infected with hepatitis C virus (HCV) genotype 1a or 1b
* HCV RNA viral load ≥10,000 IU/mL
* No prior treatment including but not limited to interferon, ribavirin, and direct-acting antivirals
* No history of cirrhosis liver biopsy within 3 years or Fibroscan® within 1 year
* Body mass index of 18 to 35 kg/m^2
* Negative for HIV and hepatitis B virus

Key Exclusion Criteria:

* Evidence of decompensated liver disease
* Evidence of medical condition other than HCV contributing to chronic liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (84):
- United States (25):
  - The Kirklin Clinic, Birmingham, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Va Long Beach Healthcare System, Long Beach, California
  - Medical Associates Research Group, San Diego, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - Orlando Immunology Center, Orlando, Florida
  - Atlanta Medical Center, Atlanta, Georgia
  - Gastrointestinal Specialists Of Georgia, Marietta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University Of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Lutherville, Maryland
  - Minnesota Gastroenterology, P.A., Saint Paul, Minnesota
  - Saint Louis University Gastroenterology & Hepatology, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - University Of North Carolina At Chapel Hill School Of Med, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor College Of Medicine, Houston, Texas
  - Research Specialists Of Texas, Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
- Argentina (3):
  - Local Institution, Ciudad de Buenos Aires, Buenos Aires
  - Local Institution, Prov. Buenos Aires, Buenos Aires
  - Local Institution, Prov de Santa Fe, Santa Fe Province
- Australia (7):
  - Local Institution, Camperdown, New South Wales
  - Local Institution, Penrith, New South Wales
  - Local Institution, Westmead Nsw, New South Wales
  - Local Institution, Greenslopes Qld, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Fitzroy, Victoria
  - Local Institution, Prahran, Victoria
- Austria (2):
  - Local Institution, Linz
  - Local Institution, Vienna
- Local Institution, São Paulo, São Paulo, Brazil
- Canada (6):
  - Local Institution, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Ottawa, Ontario
  - Local Institution, Toronto, Ontario
- Denmark (2):
  - Local Institution, Hvidovre
  - Local Institution, Odense
- France (7):
  - Local Institution, Besançon
  - Local Institution, Bondy
  - Local Institution, Grenoble
  - Local Institution, Lille
  - Local Institution, Paris
  - Local Institution, Pessac
  - Local Institution, Strasbourg
- Germany (7):
  - Local Institution, Berlin
  - Local Institution, Cologne
  - Local Institution, Essen
  - Local Institution, Frankfurt
  - Local Institution, Freiburg im Breisgau
  - Local Institution, Hamburg
  - Local Institution, Hanover
- Israel (4):
  - Local Institution, Haifa
  - Local Institution, Nazareth
  - Local Institution, Safed
  - Local Institution, Tel Aviv
- Italy (5):
  - Local Institution, Bergamo
  - Local Institution, Cisanello (pisa)
  - Local Institution, Florence
  - Local Institution, Napoli
  - Local Institution, Torino
- Poland (6):
  - Local Institution, Bialystok
  - Local Institution, Chorzów
  - Local Institution, Kielce
  - Local Institution, Mysłowice
  - Local Institution, Racibórz
  - Local Institution, Wroclaw
- Local Institution, Moscow, Russia
- Spain (3):
  - Local Institution, Alcorcón
  - Local Institution, Barcelona
  - Local Institution, Valencia
- Local Institution, Zurich, Switzerland
- United Kingdom (4):
  - Local Institution, London, Greater London
  - Local Institution, Edinburgh, Scotland
  - Local Institution, Glasgow, Scotland
  - Local Institution, Birmingham, West Midlands

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 793 participants were recruited at 90 sites in 15 countries.
Pre-assignment Details: Of the 793 participants, 605 were randomized to treatment. A total of 191 enrolled subjects did not enter the treatment period as they no longer met study entry criteria and a 602 participants were received treatment.
Groups:
- Daclatasvir + PEG-IFN Alpha-2a + Ribavirin: Participants received daclatasvir 60-mg tablet orally once daily for 24 weeks in combination with pegylated interferon alpha-2a (PEG-IFN alpha-2a)180 µg administered subcutaneously once a week for 24 or 48 weeks and ribavarin administered in a body weight stratified dose range of 1000-1200 mg per day (for participants weighing less than 75 kg, the total dose was 1000 mg per day and for those weighing greater than or equal to 75 kg, the dose was 1200 mg per day).
- Telaprevir + PEG-IFN Alpha-2a + Ribavirin: Participants received 2 telaprevir 375-mg tablets orally 3 times a day for 12 weeks. PEG-IFN alpha-2a 180 µg was coadministered subcutaneously once a week for 24 or 48 weeks depending on response, and ribavirin in a body weight stratified dose range of 1000-1200 mg per day was administered twice daily with food.
Period: Treatment
Arm/Group | Daclatasvir + PEG-IFN Alpha-2a + Ribavirin | Telaprevir + PEG-IFN Alpha-2a + Ribavirin
Started | 402 | 200
Completed | 319 | 160
Not Completed | 83 | 40
Not completed — Death | 0 | 1
Not completed — Other | 1 | 0
Not completed — Adverse Event | 25 | 25
Not completed — Lack of Efficacy | 38 | 5
Not completed — Participant withdrew consent | 1 | 2
Not completed — Poor compliance/noncompliance | 1 | 0
Not completed — Subject requested discontinue study drug | 7 | 3
Not completed — Lost to Follow-up | 9 | 4
Not completed — Participant does not meet study criteria | 1 | 0
Period: Follow-Up
Arm/Group | Daclatasvir + PEG-IFN Alpha-2a + Ribavirin | Telaprevir + PEG-IFN Alpha-2a + Ribavirin
Started | 384 (This total number includes 319 who completed treatment plus 65 who rejoined for follow-up.) | 191 (This total number includes 160 who completed treatment plus 31 who rejoined for follow-up.)
Completed | 359 | 181
Not Completed | 25 | 10
Not completed — Protocol Requires no Follow-Up | 2 | 1
Not completed — Death | 1 | 0
Not completed — Other | 4 | 2
Not completed — Participant Withdrew Consent | 6 | 1
Not completed — Lost to Follow-up | 12 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daclatasvir + PEG-IFN Alpha-2a + Ribavirin | Telaprevir + PEG-IFN Alpha-2a + Ribavirin | Total
Number analyzed (Participants) | 402 | 200 | 602
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (12.12) | 47.6 (12.29) | 46.9 (12.18)
Age, Customized [Number; unit: participants]
  Younger than 65 years | 387 | 188 | 575
  65 years and older | 15 | 12 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 81 | 226
  Male | 257 | 119 | 376

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Genotype 1b Participants With Sustained Virologic Response at Follow-up Week 12 (SVR12)
Description: SVR12 was defined as hepatitis C virus RNA levels to be lower than the limit of quantitation, ie, 25 IU/mL target detected or target not detected at follow-up Week 12.
Time Frame: Week 12 (Follow-up period)
Population: The analysis was performed in all treated participants who received at least 1 dose of active study therapy. Here, 'Number of participants analysed' signifies Genotype 1b participants assessed for SVR12 response.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Daclatasvir + PEG-IFN Alpha-2a + Ribavirin: Participants received daclatasvir 60-mg tablet orally once daily for 24 weeks in combination with pegylated interferon alpha-2a (PEG-IFN alpha-2a) 180 µg administered subcutaneously once a week for 24 or 48 weeks and ribavarin administered in a body weight stratified dose range of 1000-1200 mg per day (for participants weighing less than 75 kg, the total dose was 1000 mg per day and for those weighing greater than or equal to 75 kg, the dose was 1200 mg per day).
Arm/Group | Daclatasvir + PEG-IFN Alpha-2a + Ribavirin | Telaprevir + PEG-IFN Alpha-2a + Ribavirin
Number analyzed (Participants) | 268 | 134
Percentage of participants | 85.1 [80.2 to 89.1] | 81.3 [73.7 to 87.5]
Statistical Analysis 1: Comparison: Daclatasvir + PEG-IFN Alpha-2a + Ribavirin vs Telaprevir + PEG-IFN Alpha-2a + Ribavirin; Percentage difference between SVR12 rate in the experimental and control arms was computed using a stratum-adjusted Mantel-Haenszel confidence interval (95% level) for the difference in rates. The stratification factors were IL28B rs1297860 single nucleotide polymorphism (CC or non-CC) and baseline cirrhosis status (absent or present), unless otherwise indicated; Test type: Non-Inferiority or Equivalence — Test of noninferiority was based on noninferiority margin of -12% and 2-sided alpha level of 5%. That is, if the lower bound of the 95% CI > -12%, the Daclatasvir arm would be considered nonnferior to the telaprevir arm; Stratum-adjusted Mantel-Haenszel — Test of noninferiority carried out by taking a confidence interval (CI) for the difference in rates (daclatasvir arm minus telapravir arm). If lower bound of 95% CI difference exceeded -12%, noninferiority was demonstrated. No p-value was computed; Percentage difference = 4.3, 95% CI 2-sided [-3.3 to 11.9], Standard Deviation 3.885

2. Secondary Outcome: Percentage of Genotype 1b Participants With Rapid Virologic Response (RVR) at Week 4
Description: RVR was defined as hepatitis c virus RNA levels lower than lower limit of quantitation, ie, 25 IU/mL target not detected at Week 4 of treatment.
Time Frame: Week 4
Population: The analysis was performed in all treated participants who received at least 1 dose of active study therapy. Here, 'Number of participants analysed' signifies Genotype 1b participants assessed for RVR response.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Daclatasvir + PEG-IFN Alpha-2a + Ribavirin: Participants received daclatasvir 60-mg tablet orally once daily for 24 weeks in combination with pegylated interferon alpha-2a (PEG-IFN alpha-2a) 180 µg administered subcutaneously once a week for 24 or 48 weeks and ribavarin administered in a body weight stratified dose range of 1000 - 1200 mg per day (for participants weighing less than 75 kg, the total dose was 1000 mg per day and for those weighing greater than or equal to 75 kg, the dose was 1200 mg per day).
Arm/Group | Daclatasvir + PEG-IFN Alpha-2a + Ribavirin | Telaprevir + PEG-IFN Alpha-2a + Ribavirin
Number analyzed (Participants) | 268 | 134
Percentage of participants | 77.2 [71.7 to 82.1] | 79.1 [71.2 to 85.6]

3. Secondary Outcome: Percentage of Genotype 1b Participants With Extended Rapid Virologic Response (eRVR) at Both Week 4 and Week 12
Description: eRVR was defined as hepatitis C virus RNA levels lower than the lower limit of quantitation, ie, 25 IU/mL target not detected at both Weeks 4 and 12 of treatment.
Time Frame: Week 4, Week 12
Population: The analysis was performed in all treated participants who received at least 1 dose of active study therapy. Here, 'Number of participants analysed' signifies Genotype 1b participants assessed for eRVR response.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Telaprevir + PEG-IFN Alpha-2a + Ribavirin: Participants received 2 telaprevir 375-mg tablets orally 3 times a day for 12 weeks. PEG-IFN alpha-2a 180 µg was coadministered subcutaneously once a week for 24 or 48 weeks depending on response, and ribavirin in a body weight stratified dose range of 1000-1200mg per day was administered twice daily with food.
Arm/Group | Daclatasvir + PEG-IFN Alpha-2a + Ribavirin | Telaprevir + PEG-IFN Alpha-2a + Ribavirin
Number analyzed (Participants) | 268 | 134
Percentage of participants | 75.0 [69.4 to 80.1] | 73.1 [64.8 to 80.4]

4. Secondary Outcome: Percentage of Genotype 1b Participants With Complete Early Virologic Response (cEVR)
Description: cEVR was defined as hepatitis C virus RNA levels lower than the lower limit of quantitation, ie, 25 IU/mL target not detected at Week 12 of treatment.
Time Frame: Week 12
Population: The analysis was performed in all treated participants who received at least 1 dose of active study therapy. Here, 'Number of participants analysed' signifies Genotype 1b participants assessed for cEVR response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Daclatasvir + PEG-IFN Alpha-2a+ Ribavirin: Participants received daclatasvir 60-mg tablet orally once daily for 24 weeks in combination with pegylated interferon alpha-2a (PEG-IFN alpha-2a)180 µg administered subcutaneously once a week for 24 or 48 weeks and ribavarin administered in a body weight stratified dose range of 1000-1200 mg per day (for participants weighing less than 75 kg, the total dose was 1000 mg per day and for those weighing greater than or equal to 75 kg, the dose was 1200 mg per day).
Arm/Group | Daclatasvir + PEG-IFN Alpha-2a+ Ribavirin | Telaprevir + PEG-IFN Alpha-2a + Ribavirin
Number analyzed (Participants) | 268 | 134
percentage of participants | 90.7 [86.5 to 93.9] | 90.03 [84.0 to 94.7]

5. Secondary Outcome: Percentage of Genotype 1b Participants With Sustained Virologic Response at Follow-up Week 24 (SVR24)
Description: SVR24 was defined as hepatitis C virus RNA levels lower than the lower limit of quantitation, ie, 25 IU/mL target detected or target not detected at follow-up week 24 of treatment.
Time Frame: Week 24 (Follow-up period)
Population: The analysis was performed in all treated participants who received at least 1 dose of active study therapy. Here, 'Number of participants analysed' signifies Genotype 1b participants assessed for SVR24 response.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Daclatasvir + PEG-IFN Alpha-2a+ Ribavirin | Telaprevir + PEG-IFN Alpha-2a + Ribavirin
Number analyzed (Participants) | 268 | 134
Percentage of participants | 84.3 [79.4 to 88.5] | 80.6 [72.9 to 86.9]

6. Secondary Outcome: Percentage of Genotype 1a Participants With Sustained Virologic Response at Follow-up Week 12 (SVR12)
Description: SVR12 was defined as hepatitis C virus RNA levels lower than the lower limit of quantitation, ie, 25 IU/mL target detected or target not detected at follow-up week 12 of treatment.
Time Frame: Week 12 (Follow-up period)
Population: The analysis was performed in all treated participants who received at least 1 dose of active study therapy. Here, 'Number of participants analysed' signifies Genotype 1a participants assessed for SVR12 response.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Daclatasvir + PEG-IFN Alpha-2a + Ribavirin | Telaprevir + PEG-IFN Alpha-2a + Ribavirin
Number analyzed (Participants) | 134 | 66
Percentage of participants | 64.9 [56.2 to 73.0] | 69.7 [57.1 to 80.4]

ADVERSE EVENTS:
Arm/Group | Daclatasvir + PEG-IFN Alpha-2a + Ribavirin | Telaprevir + PEG-IFN Alpha-2a + Ribavirin
Serious Adverse Events (participants affected / at risk) | 26/402 | 20/200
Other Adverse Events (participants affected / at risk) | 384/402 | 193/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daclatasvir + PEG-IFN Alpha-2a + Ribavirin (N=402) | Telaprevir + PEG-IFN Alpha-2a + Ribavirin (N=200)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Proctitis infectious (Infections and infestations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 5
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Peritonsillar abscess (Infections and infestations) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 2
Sepsis (Infections and infestations) | 0 | 1
Bursitis infective (Infections and infestations) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Headache (Nervous system disorders) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Bipolar I disorder (Psychiatric disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 2
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Panic disorder (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daclatasvir + PEG-IFN Alpha-2a + Ribavirin (N=402) | Telaprevir + PEG-IFN Alpha-2a + Ribavirin (N=200)
Arthralgia (Musculoskeletal and connective tissue disorders) | 55 | 14
Dry skin (Skin and subcutaneous tissue disorders) | 84 | 34
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 48 | 25
Fatigue (General disorders) | 140 | 81
Myalgia (Musculoskeletal and connective tissue disorders) | 61 | 23
Pruritus (Skin and subcutaneous tissue disorders) | 107 | 75
Disturbance in attention (Nervous system disorders) | 22 | 10
Dizziness (Nervous system disorders) | 32 | 18
Insomnia (Psychiatric disorders) | 71 | 35
Pyrexia (General disorders) | 80 | 42
Rash (Skin and subcutaneous tissue disorders) | 93 | 69
Chills (General disorders) | 31 | 18
Diarrhoea (Gastrointestinal disorders) | 63 | 35
Influenza like illness (General disorders) | 85 | 38
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 11
Vertigo (Ear and labyrinth disorders) | 18 | 12
Vomiting (Gastrointestinal disorders) | 26 | 23
Abdominal pain upper (Gastrointestinal disorders) | 24 | 15
Anaemia (Blood and lymphatic system disorders) | 96 | 98
Anorectal discomfort (Gastrointestinal disorders) | 3 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 76 | 31
Nausea (Gastrointestinal disorders) | 88 | 74
Neutropenia (Blood and lymphatic system disorders) | 87 | 27
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 22 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 19 | 14
Urinary tract infection (Infections and infestations) | 7 | 10
Alopecia (Skin and subcutaneous tissue disorders) | 86 | 32
Anxiety (Psychiatric disorders) | 10 | 16
Dysgeusia (Nervous system disorders) | 23 | 21
Erythema (Skin and subcutaneous tissue disorders) | 16 | 10
Haemorrhoids (Gastrointestinal disorders) | 7 | 11
Headache (Nervous system disorders) | 137 | 57
Injection site erythema (General disorders) | 21 | 7
Injection site reaction (General disorders) | 22 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 27 | 14
Decreased appetite (Metabolism and nutrition disorders) | 61 | 39
Dyspepsia (Gastrointestinal disorders) | 17 | 16
Anal pruritus (Gastrointestinal disorders) | 3 | 25
Irritability (Psychiatric disorders) | 43 | 27
Proctalgia (Gastrointestinal disorders) | 2 | 11
Asthenia (General disorders) | 109 | 53
Depression (Psychiatric disorders) | 29 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.